CLINICAL TRIAL: NCT02720497
Title: The Efficacy of 90-Minute Versus 60-Minute Sessions of Prolonged Exposure for PTSD: A Randomized Controlled Trial in Active Duty Military Personnel
Brief Title: The Efficacy of 90-Minute Versus 60-Minute Sessions of Prolonged Exposure for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Medical University of South Carolina (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-15-1-0555
Record Dates: First submitted 2016-03-10; First posted 2016-03-28 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Posttraumatic Stress Disorder; Combat Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 60-minute Prolonged Exposure (Experimental): This treatment condition is a modified version of Prolonged Exposure therapy for PTSD. It consists of weekly weekly 60-minute sessions, with 20 minutes imaginal exposure.
  Interventions: Behavioral: 60-minute Prolonged Exposure Therapy
- 90-minute Prolonged Exposure (Active Comparator): Prolonged Exposure Therapy for PTSD consists of weekly 90-minute sessions, with 40 minutes imaginal exposure.
  Interventions: Behavioral: 90-minute Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: 60-minute Prolonged Exposure Therapy — This treatment condition is a modified version of Prolonged Exposure therapy for PTSD. It consists of weekly weekly 60-minute sessions, with 20 minutes imaginal exposure.
  Arms: 60-minute Prolonged Exposure
Behavioral: 90-minute Prolonged Exposure Therapy — Prolonged Exposure Therapy for PTSD consists of weekly 90-minute sessions, with 40 minutes imaginal exposure.
  Arms: 90-minute Prolonged Exposure

SUMMARY:
Objectives and Rationale: With up to 20% of U.S. service members returning from Iraq and Afghanistan with PTSD symptoms, a critical need exists for treatments that are both effective and efficient, enabling the greatest number possible to be treated to remission. As a highly efficacious treatment and the one with the most scientific support, Prolonged Exposure (PE) is recommended by the Institute of Medicine and being rolled out by the Departments of Defense and Veterans Affairs to help heal our war fighters' psychological wounds. A major barrier to that roll-out, however, is that PE is typically delivered in 90-minute sessions. This is difficult for military mental health providers, who because of large patient loads and pressure to see as many patients per day as possible, limit therapy sessions to 60 minutes. The primary aim of this randomized clinical trial is to determine whether PE sessions can be reduced to 60 minutes without compromising the treatment's high success rate. Preliminary evidence suggests that patients may greatly benefit from PE even when the time spent recalling and recounting the trauma memories during sessions (a key procedure called imaginal exposure) is shortened to fit into a 60-minute session. To test this hypothesis, the trial will enroll 160 San Antonio-area active duty service members who will be randomly assigned to receive PE treatment with 60- or 90-minute sessions. In an additional effort to learn more about how PE helps patients recover - and thereby gain insights to further enhance treatment benefit - the study investigators will examine what causes reductions in PTSD symptoms during PE by examining self-reported and physiological markers (e.g., heart rate reactivity) between the two treatment groups.

Research Applicability and Impact: If PE can be shown to maintain high success rates with shorter sessions, more military clinicians could offer this powerful therapy, as it would fit within time constraints of their heavy workload. This would potentially help thousands of our nation's warriors recover from the devastating psychological effects of PTSD and maintain their military careers, heal hurting relationships, and reengage in meaningful life activities. This study would further benefit the military and the general public by enhancing the readiness of our Armed Forces and reducing the public cost of service members' lost work time or veterans' disability benefits. Overloaded VA providers and even civilian therapists, who often limit sessions to 60 minutes due to insurance reimbursement requirements, may also be more likely to utilize the shorter treatment format, increasing access to evidence-base care for veterans and civilians. In addition, insights from the study's examination of biomarkers and underlying mechanisms of PE could be used to enhance care for service members, veterans, and the general public. Study risks are minimal, as a small proportion of patients may see temporary symptom increases as they deal with traumatic memories, but this is part of the recovery process. Patients receiving the shorter treatment sessions potentially may realize a lower level of treatment benefits, but preliminary evidence suggests there is good reason to believe their treatment will be equally as successful as those receiving traditional PE.

ELIGIBILITY:
Inclusion Criteria

1. Adult male and female active duty military personnel who have deployed since 9/11, ages 18-65 seeking treatment for Posttraumatic Stress Disorder (PTSD).
2. Either diagnosis of PTSD as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview, OR, CAPS-5 severity ≥ 25 and a PCL-5 score of ≥ 25.
3. Able to speak, read, and write English.

Exclusion Criteria

1. Current manic or psychotic symptoms required immediate stabilization or hospitalization (as determined by the Manic and Psychosis sections of the Mini International Neuropsychiatric Interview; MINI)
2. Current severe alcohol use symptoms (as determined by a score of ≥ 4 on items #4-6 and a total score of ≥ 20 on the Alcohol Use Disorders Identification Test; AUDIT).
3. Evidence of a severe traumatic brain injury as determined by marked impairment in communication or comprehension.
4. Current suicidal ideation severe enough to warrant immediate crisis intervention (as determined by the Depressive Symptoms Index-Suicidality Subscale and corroborated by a clinical risk assessment by a credentialed provider).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Interviewer-assessed Posttraumatic Stress Disorder (PTSD) symptoms as measured by the Clinician Administered PTSD Scale for Diagnostic Statistical Manual (DSM)-5 | Change from baseline to 1-month follow-up (post-treatment)

SECONDARY OUTCOMES:
Self-reported Posttraumatic Stress Disorder (PTSD) symptoms Posttraumatic Stress Checklist for Diagnostic Statistical Manual (DSM)-5 | Change from baseline to 1-month follow-up (post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Edna Foa, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided